CLINICAL TRIAL: NCT00782977
Title: Oxygenation Via Nasal Cannulae Prevents Arterial Hypoxemia During the Apneic Period in Paralyzed Patients
Brief Title: Apneic Oxygenation Via Nasal Cannulae Prevents Arterial Hypoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Dr Chris Christodoulou, Dept. of Anesthesia and Perioperative Medicine, St. Boniface General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2008:129
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2011-05

CONDITIONS: Hypoxia
Keywords: Apneic oxygenation; Apneic diffusion oxygenation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Sham Comparator): Nasal cannulae with no oxygen flow
  Interventions: Other: Nasal oxygen therapy
- 2 (Active Comparator): Nasal cannulae with oxygen flow at 5 L/minute
  Interventions: Other: Nasal oxygen therapy
- 3 (Active Comparator): Nasal cannulae with oxygen flow at 10 L/minute
  Interventions: Other: Nasal oxygen therapy

INTERVENTIONS:
Other: Nasal oxygen therapy — Arm 1: Nasal cannulae with no oxygen flow. Arm 2: Nasal cannulae with oxygen flow at 5 L/min Arm 3: Nasal cannulae with oxygen flow at 10 L/min

SUMMARY:
The purpose of the study is to evaluate the effectiveness of continuous oxygen provided by nasal prongs in preventing or delaying hypoxemia during the apneic period that occurs after induction of general anesthesia. This will be evaluated by measuring the arterial oxygen tension (PaO2).

The study will also evaluate whether there is any difference in PaO2 when using nasal prongs with flow rates of 5 L/minute versus 10 L/minute of oxygen.

DETAILED DESCRIPTION:
Certain patient populations are at risk for rapid desaturation and the rapid development of hypoxemia (eg. morbidly obese and pregnant patients). Using pulse oximetry, it has already been shown that oxygen provided with a catheter inserted into the nasopharynx is effective in delaying the desaturation that occurs with apnea before the trachea is intubated. It has also been shown that apneic oxygenation with nasal prongs at 5 L/min during fibreoptic intubation can delay the onset of hypoxemia.

The study will evaluate whether there is any significant difference in the PaO2 (arterial oxygen tension, as measured by an arterial blood gas) when nasal prongs are used to provide apneic oxygenation in paralyzed patients at flows of 5 L/min compared to 10 L/min.

The study aims to demonstrate that apneic oxygenation using nasal prongs is effective in preventing or delaying hypoxemia (by measuring PaO2), and that this technique may be used to prevent morbidity and mortality in all clinical areas (not only in the Operating Room environment) where airway management is undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females
2. ASA Class 1-3
3. Ages of 18 to 65
4. Elective surgery under general anesthesia
5. No evidence of significant cardiac, respiratory or gastrointestinal disease
6. No contraindications to the insertion of a radial arterial catheter

Exclusion Criteria:

1. Evidence of a difficult airway (expected difficult intubation identified from patient history or clinical examination)
2. Features suggestive of difficult bag mask ventilation
3. Significant GERD requiring medical therapy
4. Significant respiratory disease (including severe asthma or COPD, oxygen dependency, pulmonary hypertension)
5. Significant cardiac disease (ischemic heart disease, severe aortic and mitral stenosis and/or regurgitation, EF < 50% if known)
6. Inability to lie flat (skeletal deformities, orthopnea, congestive cardiac failure)
7. PaO2 < 200 mmHg on ABG after adequate preoxygenation to an ETO2 > 85%
8. Hemoglobin < 100 g/L
9. BMI > 40 kg/ m2
10. Pregnancy
11. Patient unwillingness or refusal to participate
12. Inability to consent (dementia) or cooperate (mentally challenged)
13. Inability to communicate well or to understand English (language barrier, dysphasia)
14. Neuromuscular disorders
15. Known or presumed cervical spine instability (cervical spine fractures, rheumatoid arthritis)
16. Patients undergoing neurosurgical procedures
17. Any clinical or radiological evidence of increase in intracranial pressure
18. Any requirement for rapid sequence intubation
19. Inability to tolerate the apneic period
20. Allergy to any of the agents used for induction of general anesthesia in the study
21. Arterial insufficiency with poor collateral circulation to the hand (tested with Doppler ultrasound or clinically by palpation with the Allen test)
22. Inability to cannulate an artery for monitoring and sampling purposes
23. Uncorrected coagulopathy
24. Baseline hypercarbia (PaCO2 > 50 mmHg)
25. Known or suspected obstructive sleep apnea
26. Significant nasal obstruction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
PaO2 in mmHg (arterial oxygen tension as measured by an arterial blood gas) | Arterial blood gases taken at one minute intervals post induction in the apneic period, for a total of 4 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Chris Christodoulou, MBChB, FRCPC, Principal Investigator — Dept of Anesthesia and Perioperative Medicine, St. Boniface General Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada